CLINICAL TRIAL: NCT06321926
Title: Evaluation of the "ActiveWaiting App" Encouraging Active Exercise-related Use of Waiting Time. A Waitlist Control Study
Brief Title: Evaluation of the "ActiveWaiting App" Encouraging Active Exercise-related Use of Waiting Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Institute for Digital Health and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 154/2023
Record Dates: First submitted 2024-02-27; First posted 2024-03-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity
Keywords: sedentary behaviour; behaviour change; digital health
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the intervention group or the waitlist control group. The intervention group uses the ActiveWaiting App for a week, the waitlist control group starts with a control period (one week), before using the App for a week.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcomes will be selected via lime survey. Allocation to the groups will be concealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group use the ActiveWaiting App for one week.
  Interventions: Device: ActiveWaiting App
- Waitlist control group (Other): Participants in the waitlist control group go through a one-week control period without any intervention first, before they are using the app for one week.
  Interventions: Device: ActiveWaiting App

INTERVENTIONS:
Device: ActiveWaiting App — The final prototype aims at increasing physical activity during the day by providing exercises for waiting periods and other idle time periods. The user can choose from a pool of exercises from five different categories (11 exercises for endurance, 65 exercises for strength, 67 exercises for flexibility, 11 exercises for relaxation, or 5 exercises for balance). Additionally, within each category, the user can choose only "discrete" exercises which are not noticeable to an observer. If the user has used the app before, the last or previously saved settings can be chosen. Every input field has an information icon showing a short description of the input field.

SUMMARY:
The goal of this study (waitlist control study) is to evaluate the effectiveness of the ActiveWaiting App on increasing physical activity and improving quality of life in physically inactive adults in Austria.

The main questions it aims to answer are:

1. Does the provision of the ActiveWaiting App lead to increased physical activity behaviour, compared to a no-intervention control group?
2. Does the provision of the ActiveWaiting App lead to increased health-related quality of life, compared to a no-intervention control group? Participants will use the ActiveWaiting App over a period of seven days. During this period, they will answer daily questionnaires (3 - 6 questions) in order to gather their actual physical activity behaviour. Before and after the intervention period additional questionnaires on health-related quality of life will be sent to the participants.

Participants in the waitlist control group will have a control period (seven days) before using the app.

Researchers will compare the intervention group with the waitlist control group to see if the ActiveWating App has an effect

* on physical activity behaviour and
* on quality of life.

DETAILED DESCRIPTION:
A randomized waitlist control design will be chosen to answer the research question. Participants will be randomly assigned to the intervention group or to the waitlist control group. Block randomization with permutated block sizes will ensure that both study arms are recruited evenly over time. Allocation to the groups will be concealed. The waitlist control group will have the opportunity to use the ActiveWaiting App after the control period. Intervention and control period will be 1 week. Demographic data will be collected before randomization.

Additionally to the primary research questions, the following research questions will be addressed for explorative purposes:

* How much is the ActiveWaiting App used for active waiting and breaking time?
* Which category of exercises are used for this purpose?

ELIGIBILITY:
Inclusion Criteria:

* a sedentary lifestyle (expressed in a full to part-time sedentary job)
* using a smart phone seven days a week
* ability to operate an app on the smart phone
* age between 18 and 65 years

Exclusion Criteria:

* prior usage of the ActiveWaiting App
* achieving the World Health Organization (WHO) recommendations for physical activity (assessed via Rapid Assessment of physical Activity RAPA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Amount of physical activity in minutes per day | up to 2 weeks
  Participants are asked to report their physical activity twice a day (noon and evening).
EQ VAS / EQ-5D-5L | up to 2 weeks
  The EQ VAS (EuroQol Visual Analog Scale) is the last item in the EQ-5D-5L (EuroQol - 5 Dimension - 5 Level) Questionnaire. It records the respondent's overall current health on a visual analogue scale. The endpoints are labelled as 'The best health you can imagine' (=100) and 'The worst health you can imagine' (=0). The EQ VAS provides a quantitative measure of the person's perception of their overall health and is used in this study.

SECONDARY OUTCOMES:
App usage - exercise session length | 7 days
  Exercise session length will be recorded in seconds and is defined by the time spent in each category (endurance, strength, balance, flexicility and relaxation) of provided exercises.
App usage - total duration per session | 7 days
  The duration of each session will be recorded in seconds, based on the time spent with exercises, regardless of the category.

CONTACTS AND LOCATIONS:
Locations (1):
- FH Campus Wien, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No